CLINICAL TRIAL: NCT04157114
Title: A Double-Blind, Randomized, Controlled Trial of MAP4343 Treatment, a Ligand of the Neurospecific Microtubule Associated Protein-2, for Alcohol Use Disorder
Brief Title: MAP4343 Treatment for Alcohol Use Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The FDA requested Mapreg conduct an alcohol interaction study which was not feasible due to the COVID-19 pandemic.
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Mapreg (Industry)
Responsible Party: Principal Investigator, Barbara J. Mason, Principal Investigator, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAP2019; P60AA006420 (NIH)
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol-Related Disorders; Substance-Related Disorders; MAP4343; Alcohol Treatment; Alcohol
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAP4343 (Active Comparator): Subjects will receive daily oral doses of MAP4343 for 6 weeks in conjunction with 6 weeks of manual-guided counseling
  Interventions: Drug: MAP4343; Behavioral: Standardized behavioral counseling
- Placebo (Placebo Comparator): Subjects will receive matched placebo for 6 weeks in conjunction with 6 weeks of manual-guided counseling
  Interventions: Drug: Placebo; Behavioral: Standardized behavioral counseling

INTERVENTIONS:
Drug: MAP4343 — Subjects will receive daily oral doses of MAP4343 for 6 weeks in conjunction with 6 weeks of manual-guided counseling
  Arms: MAP4343
Drug: Placebo — Subjects receive matched placebo for 6 weeks in conjunction with 6 weeks of manual-guided counseling
  Arms: Placebo
Behavioral: Standardized behavioral counseling — Subjects receive manually-guided counseling 1 time per week for a 6 week duration
  Other Names: Manually-guided therapy

SUMMARY:
This is a Phase 2, single-site, randomized, double-blind, placebo-controlled, proof-of-concept (POC) study involving 6 weeks of MAP4343 in conjunction with 6 weeks of manual-guided counseling, with 2 follow-up visits at 1 week and 1 month post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers, 18-65 years of age
2. Meets Diagnostic and Statistical Manual (DSM)-5 criteria for current Alcohol Use Disorder (AUD) of moderate or greater severity, defined by DSM-5 as ≥ 4 symptoms
3. In the month prior to screening, reports drinking ≥ 21 standard drinks per week if male, ≥ 14 if female, with at least one heavy drinking day (males: ≥ 5 drinks, females: ≥ 4 drinks) per week
4. Seeking research-based outpatient treatment for AUD and willing to comply with the protocol, take daily oral medication for 6 weeks and complete 10 study visits
5. Abstinent a minimum of 3 days (but not more than 30 days) prior to randomization
6. Negative Blood Alcohol Concentration (BAC) and a Clinical Institute Withdrawal Assessment (CIWA) score of ≤ 9 at randomization
7. In acceptable health in the judgment of the study physician, on the basis of interview, medical history, physical exam, electrocardiogram (ECG), urine test, and routine lab tests
8. Females with childbearing potential must have a negative pregnancy test on both the screening and randomization visits and agree to use non-hormonal effective birth control for the study duration and 1 month post treatment.
9. Subjects must be able to complete and understand questionnaires and study procedures in English and sign an informed consent

Exclusion Criteria:

1. Significant medical disorders or clinically significant findings on ECG, urine or blood tests that increase potential risk or interfere with study participation as determined by the Study Physician
2. Liver function tests more than 3 times the upper limit of normal
3. Meets DSM-5 criteria for a major Axis I disorder including mood or anxiety disorders or substance use disorders other than alcohol or nicotine use disorders or mild cannabis use disorder
4. Urine drug test positive at screening for abused drugs other than cannabis. Subjects using cannabis will be excluded if they meet criteria for cannabis use disorder ≥ moderate level of severity
5. Treatment within the month prior to screening with an investigational drug or vaccine, or drugs that may influence study outcomes, e.g., disulfiram, naltrexone, acamprosate
6. Chronic use or need for psychotropic drugs. Note: some drugs with psychotropic properties (e.g., anti-hypertensive drugs) or antidepressant medication taken at a stable dose for ≥ 3 months and no longer meeting criteria for depressive or anxiety disorders are allowed if their use is judged by both the investigator and study physician not to pose a safety risk or impact the results of the study
7. No fixed domicile and/or no availability by home or mobile telephone
8. Treatment mandated by a legal authority
9. Failure to comply with study procedures
10. Subjects who require medical detoxification (Note: Subjects may proceed with study evaluation after completion of detoxification)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Timeline Follow-Back (TLFB) Interview | 90-day period prior to and throughout the study
  The Timeline Follow-Back Interview provides quantity and frequency estimates of alcohol consumption for the 90-day period prior to and throughout the study.
Visual Analogue Scale of Craving (VAS; adapted from ACQ) | At subject's Week 2 human laboratory session
  The Visual Analogue Scale of Craving has 4 questions to assess domains of alcohol craving: the intention to drink, loss of control, relief craving, and urge intensity with a 0-20 point visual analogue scale for each item, with 0 indicating no craving and 20 indicating severe craving.

SECONDARY OUTCOMES:
Alcohol Craving Questionnaire-Short Form (ACQ-SF) | Subjects will followed for up to 10 weeks
  The Alcohol Craving Questionnaire-Short Form has 12 questions about alcohol craving which are each scored 1-7, then summed for a weekly score between 7 and 84, with higher scores indicating greater craving.
Beck Depression Inventory (BDI-II) | Subjects will be followed for up to 10 weeks
  The Beck Depression Inventory II consists of 21 questions assessing depression symptoms answered with scores between 0-3, summed for a weekly total score between 0 and 63, higher scores indicate more depression.
Pittsburgh Sleep Quality Index (PSQI) | Subjects will be followed for up to 10 weeks
  The Pittsburgh Sleep Quality Index, modified for weekly administration, consists of 9 questions about sleep habits which are answered on a scale of 0-3. Results are sorted into 7 sub scales re-scored 0-3, then sub scales are summed for a weekly total score between 0 and 21, with higher scores indicating greater sleep impairment.
State-Trait Anxiety Inventory (STAI) | Subjects will be followed for up to 10 weeks
  The State-Trait Inventory has 20 questions for assessing state anxiety and 20 for trait anxiety answered with scores between 1-4, summed for a weekly total score between 20 and 80, higher scores indicate more anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- The Scripps Research Institute Pearson Center for Alcoholism and Addiction Research, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No